CLINICAL TRIAL: NCT03628885
Title: "Keeping All Teens Healthy Study": An Evaluation of Tailored Messages to Address Parental Questions About HPV Vaccination
Brief Title: An Evaluation of Tailored Messages to Address Parental Questions About HPV Vaccination
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 1807664964
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Results first posted 2019-04-02 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2018-07

CONDITIONS: Human Papilloma Virus Vaccines; Attitude to Health

STUDY DESIGN:
Intervention Model Description: Factorial Assignment
Who Masked: Participant, Investigator
Masking Description: Intervention videos delivered via anonymous online surveys through Survey Sampling International. Randomization to condition is built into the online survey. Participants will not know to which condition they will be randomized. Investigators are blinded by virtue of the built in randomization and anonymity of the survey.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- General Vaccine Information (No Intervention): Brief (47 second) animated informational video about vaccines recommended for all young adolescents.
- Top Concern Tailored Intervention (Experimental): Intervention includes the General Vaccine Information video plus a brief (< 50 sec) animated video address the parent's top ranked question or concern from the provided list of possible concerns: 1. "I need more information about the vaccine"; 2. "My child is too young"; 3. "I am concerned about the long-term health effects or safety of the vaccine"; 4. "My child's health care provider did not recommend it or said my child could wait"; 5. "The vaccine is not required for school"; 6. "Other / none of the above". For those indicating #6, they will receive the same video as those indicating #1 (need more information).
  Interventions: Behavioral: Top Concern Tailored Intervention
- All Concerns Tailored Intervention (Experimental): Intervention includes the General Vaccine Information video plus one or more brief (< 50 sec) animated videos that address all of the parent's indicated question or concern from the provided list of possible concerns: 1. "I need more information about the vaccine"; 2. "My child is too young"; 3. "I am concerned about the long-term health effects or safety of the vaccine"; 4. "My child's health care provider did not recommend it or said my child could wait"; 5. "The vaccine is not required for school"; 6. "Other / none of the above".
  Interventions: Behavioral: All Concerns Tailored Intervention

INTERVENTIONS:
Behavioral: Top Concern Tailored Intervention — General Vaccine Information video plus a brief (< 50 sec) animated video address the parent's top ranked question or concern from the provided list of possible concerns.
  Arms: Top Concern Tailored Intervention
Behavioral: All Concerns Tailored Intervention — General Vaccine Information video plus one or more brief (< 50 sec) animated videos that address all of the parent's indicated question or concern from the provided list of possible concerns.
  Arms: All Concerns Tailored Intervention

SUMMARY:
The purpose of this study is to investigate mother's attitudes about vaccinating their 11-14 year old children against the human papillomavirus (HPV). Among mothers who do not plan to vaccinate their child, the investigators will assess the influence of brief videos tailored to mothers' questions and concerns. Mothers will be randomized to one of three arms: 1. General video message about vaccination; 2. General message plus a brief video addressing the mother's primary concern; or 3. General message plus videos address all of mother-indicated concerns. The outcome of interest is intention to vaccinate. Our hypothesis is that the tailored videos will lead to increased intention to vaccinate.

DETAILED DESCRIPTION:
Attitudes will be assessed through a Web-based survey administered by Survey Sampling International (SSI). The projected sample size is approximately 3,500, comprising mothers or female guardians of at least one child aged 11-14 who live in the United States. The survey will take no more than 20 minutes to complete. Mothers who indicate that they do not plan to vaccinate their children in the next year will be randomized to view brief videos tailored to their questions or concerns about HPV vaccination. The outcome of interest is intention to vaccinate. Mothers who have vaccinated their child or intend to vaccinate their child will be asked a separate set of questions relevant to this information.

Mothers who indicate that they do not intend to vaccinate their child against HPV will be asked about their questions or concerns regarding HPV vaccination (from a pre-populated list of common concerns). Mothers will be randomized to one of three arms: 1. A general information video; 2. The general video plus a video addressing their top concern; or 3. The general video plus one or more videos addressing all of their concerns. Each video is less than 50 seconds in length.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Lives in one of 26 US states with lower rates of HPV vaccination (New Jersey, Virginia, West Virginia, Alabama, Florida, Kentucky, Mississippi, North Carolina, South Carolina, Tennessee, Indiana, Minnesota, Ohio, Arkansas, Louisiana, New Mexico, Oklahoma, Kansas, Missouri, Montana, South Dakota, Utah, Wyoming, Idaho, Texas, Iowa)
* Mother or female legal guardian of at least one child aged 11-14 years
* Able to read and understand English
* Target child must not have received any doses of HPV vaccine
* The mother/respondent must indicate that she is not sure that she will vaccinate the target child in the next year.

Exclusion Criteria:

* Under 18 years of age
* Not a mother or female legal guardian of at least one child ages 11-14 years
* Not living in the United States or in one of the above designated states within the U.S.
* Not able to understand or read English
* Target child has already received at least 1 dose of HPV vaccine
* The mother/respondent indicates (before the intervention) that she definitely intends to vaccinate the target child with HPV vaccine in the next year.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Mothers or female guardians of children 11-14 years of age
Enrollment: 908 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2018-09-27 (Actual); Study Completion 2018-09-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory D Zimet, PhD, Principal Investigator — Indiana University
Locations (1):
- Indiana University, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Srivastava T, Head KJ, O'Dell SM, Feemster KA, Panozzo CA, Zimet GD, Kornides ML. Characterizing U.S. mothers with high human papillomavirus vaccine intent yet unvaccinated adolescents. Prev Med. 2023 Apr;169:107472. doi: 10.1016/j.ypmed.2023.107472. Epub 2023 Feb 26. PMID 36854366
- [Derived] Panozzo CA, Head KJ, Kornides ML, Feemster KA, Zimet GD. Tailored Messages Addressing Human Papillomavirus Vaccination Concerns Improves Behavioral Intent Among Mothers: A Randomized Controlled Trial. J Adolesc Health. 2020 Aug;67(2):253-261. doi: 10.1016/j.jadohealth.2020.01.024. Epub 2020 Mar 18. PMID 32199723

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | General Vaccine Information | Top Concern Tailored Intervention | All Concerns Tailored Intervention
Started | 306 | 299 | 303
Completed | 267 | 252 | 243
Not Completed | 39 | 47 | 60

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | General Vaccine Information | Top Concern Tailored Intervention | All Concerns Tailored Intervention | Total
Number analyzed (Participants) | 306 | 299 | 303 | 908
Age, Customized [Count of Participants; unit: Participants]
  21-25 years old | 0 | 1 | 1 | 2
  25-30 years old | 15 | 13 | 12 | 40
  31-35 years old | 72 | 64 | 55 | 191
  36-40 years old | 84 | 72 | 67 | 223
  41-45 years old | 63 | 75 | 70 | 208
  46-50 years old | 39 | 38 | 41 | 118
  51-55 years old | 16 | 16 | 23 | 55
  56-60 years old | 5 | 5 | 11 | 21
  61-65 years old | 2 | 3 | 1 | 6
  66-70 years old | 2 | 2 | 1 | 5
  70-75 years old | 0 | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female: Female | 306 | 299 | 303 | 908
  Female: Male | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 217 | 225 | 233 | 675
  Non-Hispanic Black | 31 | 16 | 20 | 67
  Non-Hispanic Other | 28 | 33 | 37 | 98
  Hispanic | 30 | 25 | 13 | 68
Child's Sex: Female, Male [Count of Participants; unit: Participants]
  Females | 153 | 152 | 155 | 460
  Males | 153 | 147 | 148 | 448
Child's Age, Continuous [Mean (Standard Deviation); unit: Years] | 12.28 (1.12) | 12.33 (1.15) | 12.60 (1.15) | 12.40 (1.15)

OUTCOME MEASURES:

1. Primary Outcome: Intention to Vaccinate Against HPV in the Next 12 Months
Description: Each parent will be asked to respond to this question. The response will be scaled from 1-10 in terms of parental intent regarding vaccination, with higher scores meaning greater parental intent to vaccinate children.
Time Frame: Immediately after video intervention has been administered
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | General Vaccine Information | Top Concern Tailored Intervention | All Concerns Tailored Intervention
Number analyzed (Participants) | 267 | 252 | 243
score on a scale | 3.49 [3.2 to 3.8] | 3.87 [3.6 to 4.2] | 4.16 [3.8 to 4.6]
Statistical Analysis 1: Comparison: General Vaccine Information vs Top Concern Tailored Intervention vs All Concerns Tailored Intervention; Test type: Superiority; p < .02, ANOVA — Adjusted for mother's educational level, which differed across groups. A priori threshold for statistical significance = P<.05
Statistical Analysis 2: Comparison: General Vaccine Information vs Top Concern Tailored Intervention; Test type: Superiority; p = .07, ANOVA — [p-value comment as in outcome 1, analysis 1]
Statistical Analysis 3: Comparison: General Vaccine Information vs All Concerns Tailored Intervention; Adjusted for mother's educational level, which differed across groups. A priori threshold for statistical significance = P<.05; Test type: Superiority; p < .01, ANOVA — [p-value comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: 20 minutes
Description: This study involved participants completing a 20 minute online survey. Therefore, there was zero risk for either mortality or serious adverse events.
Arm/Group | General Vaccine Information | Top Concern Tailored Intervention | All Concerns Tailored Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/306 | 0/299 | 0/303

LIMITATIONS AND CAVEATS:
A limitation of this trial is that the outcome is intention to vaccinate, rather than actual vaccination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/85/NCT03628885/Prot_SAP_000.pdf